CLINICAL TRIAL: NCT07022912
Title: Objective Assessment of Gastrointestinal Involvement in Patients With Systemic Sclerosis and Gastroesophageal Reflux Symptoms Refractory to Proton Pump Inhibitors.
Brief Title: PPI Refractory - GERD Mechanisms in Systemic Sclerosis
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)185/2025
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Systemic Sclerosis (SSc); GERD (Gastroesophageal Reflux Disease)
Keywords: GERD mechanisms; gastrointestinal involvement; systemic sclerosis
MeSH Terms: conditions — Scleroderma, Systemic; Gastroesophageal Reflux | interventions — Postprandial Period; Ethanol; Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with SSc and PPI-refractory GERD symptoms: Study Subjects:
  Patients will be recruited from the outpatient clinics of the Autoimmune Diseases Unit or the Gastroenterology Department at the Vall d'Hebron University Hospital (HUVH), Barcelona.
  Inclusion Criteria:
  Diagnosis of systemic sclerosis according to the 2013 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria and/or LeRoy criteria.
  Age ≥ 18 years.
  Presence of gastroesophageal reflux symptoms, defined as heartburn and/or regurgitation occurring at least three times per week over the past three months, despite ongoing treatment with PPIs.
  Interventions: Other: educational healthcare intervention; Diagnostic Test: Objective assessment of GI motility; Diagnostic Test: Evaluation of GERD severity

INTERVENTIONS:
Other: educational healthcare intervention — This intervention will be applyed at the beginning of the study
  Other Names: avoiding late dinners; not lying down for at least 2 hours after meals; avoiding tobacco and alcohol; avoiding large or high-fat meals
Diagnostic Test: Objective assessment of GI motility — Objetive assessment of gastrointestinal dysmotility in GI organs (esophagus, stomach, small bowel) will be performed using state of the art tests.
  Other Names: Gastric emptying test; Small bowel manometry; High-resolution esophageal manometry; Abdominal CT scan
Diagnostic Test: Evaluation of GERD severity — Objective evaluation of GERD severity on PPI therapy will be performed.
  Other Names: upper GI endoscopy (on PPI); pH-impedance monitoring (on PPI)

SUMMARY:
The goal of this observational study is to learn about the mechanisms of gastroesophageal reflux disease (GERD) in patients with systemic sclerosis (SSc) who continue to experience reflux symptoms despite treatment with proton pump inhibitors (PPIs). The main question it aims to answer is:

What are the underlying gastrointestinal mechanisms contributing to PPI-refractory reflux symptoms in patients with SSc?

Participants with a confirmed diagnosis of SSc and persistent reflux symptoms despite PPI therapy will undergo standard-of-care diagnostic tests, including high-resolution esophageal manometry and pH-impedance monitoring. Clinical data and test results will be collected and analyzed to identify patterns of motility dysfunction and reflux characteristics associated with refractory symptoms.

DETAILED DESCRIPTION:
Background:

Gastroesophageal reflux disease (GERD) is one of the most frequent gastrointestinal manifestations in patients with systemic sclerosis (SSc). However, a significant proportion of these patients experience symptoms that are refractory to treatment with proton pump inhibitors (PPIs), suggesting the involvement of underlying pathophysiological mechanisms that are not yet fully defined. Motor dysfunction in other segments of the gastrointestinal tract may contribute to this refractoriness, but studies addressing this in the SSc population have been limited. Currently, there are no personalized diagnostic algorithms that integrate symptoms, objective motility findings, and clinical characteristics in patients with SSc and GERD. Our goal is to identify the mechanisms associated with the severity of PPI-refractory GERD in SSc and to develop a practical and cost-effective diagnostic model based on objective data to enable personalized medicine.

Hypothesis:

PPI-refractory GERD in patients with systemic sclerosis can be assessed more sensitively and accurately through objective evaluation of motility across different gastrointestinal organs.

Objective:

To assess the pathophysiological mechanisms associated with the severity of refractory GERD in patients with SSc using objective motility tests and clinical markers, and to develop a diagnostic algorithm to guide personalized treatment based on the organ affected.

Methods:

This is a prospective clinical cohort study. Patients with SSc and symptoms of GERD refractory to PPIs will be included. Clinical, immunological, and demographic variables will be collected. Esophageal symptoms and quality-of-life impact will be assessed using validated questionnaires. Advanced gastrointestinal motility tests (gastric emptying scintigraphy and high-resolution intestinal manometry) will be performed to evaluate mechanisms associated with reflux severity (presence of erosive esophagitis and esophageal acid exposure).

Relevance:

This study addresses a common clinical challenge in patients with SSc: the persistence of GERD symptoms despite acid-suppressive treatment with PPIs. This project proposes to elucidate the pathophysiological mechanisms associated with GERD severity using motility tests available in clinical practice, and to develop a personalized approach based on objective motility assessment. This will allow the identification of the underlying mechanisms of treatment-refractory GERD and, in the future, the evaluation of targeted therapies addressing the associated dysmotility. The development of a diagnostic algorithm will support clinical decision-making, promote rational use of invasive tests, and optimize patient management, with a potential impact on improving quality of life and healthcare efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Systemic sclerosis by ACR/EULAR 2023 criteria AND/OR Leroy Medsger classification criteria
* Reflux symptoms (Heartburn AND/OR Regurgitation), at least 3 times a week over the last 3 months despite PPI therapy

Exclusion Criteria:

* Previous surgery altering the anatomy or motility of the upper digestive tract, including fundoplication, esophageal myotomy, gastrectomy, or bariatric surgery.

Severe pulmonary or cardiac disease requiring intravenous vasodilators, continuous oxygen therapy, or ventricular assist devices, preventing the performance of gastrointestinal motility tests.

Pregnancy at the time of evaluation or planned pregnancy during the duration of the study.

Neuromuscular disorders other than systemic sclerosis that may affect gastrointestinal motility.

Prior diagnosis of functional gastrointestinal disorders, such as irritable bowel syndrome or functional dyspepsia, that may interfere with the interpretation of results.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with systemic sclerosis and PPI-refractory reflux symptoms who are members of the Spanish Association of Patients with Systemic Sclerosis and/or those recruited from outpatient clinics at participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of PPI-refractory GERD | At the end of double PPI and health intervention period (8 - 12 weeks)
  The presence of erosive esophagitis B,C, or D on endoscopy, acid exposure time > 4% or > 80 reflux episodes, as per Lyon 2.0 criteria, will be considered refractory GERD.

SECONDARY OUTCOMES:
Gastrointestinal dysmotility associations | After 8 weeks on double PPI therapy, during week 8 to 12.
  prevalence of delayed gastric emptying, esophageal dysmotility and small bowel dysmotility.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alcala-Gonzalez LG, Guillen-Del-Castillo A, Aguilar A, Barber C, Codina C, Marin Garcia A, Malagelada C, Simeon-Aznar CP. Impact of gastrointestinal symptoms and psychological distress on quality of life in systemic sclerosis: a cross-sectional study. BMJ Open. 2024 Nov 27;14(11):e089725. doi: 10.1136/bmjopen-2024-089725. PMID 39609018
- [Background] Alcala-Gonzalez LG, Guillen-Del-Castillo A, Aguilar Cayuelas A, Barber Caselles C, Codina-Clavaguera C, Marin Garcia A, Serra J, Malagelada C, Simeon-Aznar CP. Gastrointestinal dysmotility is associated with proton pump inhibitor refractory oesophagitis in patients with systemic sclerosis. Rheumatology (Oxford). 2025 May 1;64(5):3074-3079. doi: 10.1093/rheumatology/keae481. PMID 39250735